CLINICAL TRIAL: NCT01441882
Title: A Phase II Study of Dasatinib in Chronic Lymphocytic Leukemia in Patients Who Exhibit in Vitro Dasatinib Sensitivity
Brief Title: Dasatinib in Treating Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Stephen Spurgeon, Associate Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006146; NCI-2011-03136 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEM 10010-L; OHSU-6146; BMS CA180-280; IRB00006146 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2011-09-21; First posted 2011-09-28 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Refractory Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dasatinib) (Experimental): Patients receive dasatinib PO QD during course 1 and if tolerated, BID in subsequent courses. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well dasatinib works in treating patients with chronic lymphocytic leukemia (CLL). Dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the biologic target activity of dasatinib in CLL patients found to have pre-treatment in vitro dasatinib cytotoxicity (as defined by a >= 50% decrease in absolute lymphocyte count and/or bone marrow CLL count and/or lymph node or spleen size).

SECONDARY OBJECTIVES:

I. To evaluate overall objective response rates per CLL National Cancer Institute (NCI) working group.

II. To determine drug safety and tolerability of dasatinib in patients with CLL.

III. To determine overall (OS) and progression-free survival (PFS).

TERTIARY OBJECTIVES:

I. To determine if v-src avian sarcoma (Schmidt-Ruppin A-2) viral oncogene homolog (SRC), Bruton agammaglobulinemia tyrosine kinase (BTK), or tec protein tyrosine kinase (TEC) family kinase inhibition correlates with clinical response.

II. To determine which prognostic subgroups (presence of >= 1 of the following: 11q or 17p deletion; cluster of differentiation [CD]38 or zeta-chain-associated protein kinase 70 [Zap 70] expression; unmutated immunoglobulin heavy chain [IgVH]) respond to dasatinib therapy.

III. To evaluate differences in baseline CLL gene expression between CLL samples that are sensitive or in-sensitive to dasatinib.

IV. To analyze changes in CLL gene expression after dasatinib treatment. V. To evaluate dasatinib pharmacokinetics. VI. To evaluate changes in type I receptor tyrosine kinase-like orphan receptor (ROR-1) expression with dasatinib treatment.

VII. To correlate response to pre-clinical IC50 in the presence/absence of HS-5 conditioned media.

VIII. To explore role of possible kinase mutations related to dasatinib response.

IX. To measure chemokines before and during treatment.

OUTLINE:

Patients receive dasatinib orally (PO) once daily (QD) during course 1 and if tolerated, twice daily (BID) in subsequent courses. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal information
* Eastern Cooperative Oncology Group (ECOG) =< 2
* In vitro dasatinib sensitivity (IC 50 =< 50 nm per MTS assay)
* Diagnosis of CLL and must meet one of the following:

  * Relapsed CLL in all patients who have failed at least one prior treatment, regardless of risk group
  * OR De novo (treatment-naïve) patients age >= 65 who are not candidates for or do not want to pursue aggressive chemotherapy treatment
* Have indications for treatment or evidence of progressive disease defined as follows (1996 NCI working group):

  * Massive or progressive splenomegaly
  * Massive lymph nodes (>= 10 cm), nodal clusters (>= 10 cm), or progressive lymphadenopathy
  * Symptomatic anemia and/or thrombocytopenia (Rai stages III or IV disease)
  * Autoimmune hemolytic anemia and/or thrombocytopenia that are poorly responsive to corticosteroid therapy
  * Progressive lymphocytosis with increase in lymphocyte count of >= 50% over a 2-month period or an anticipated doubling time of < 6 months
  * Repeated episodes of infection
* Have not received CLL treatment within the past 2 weeks
* Total bilirubin < 2.0 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 2.5 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN
* Serum creatinine < 2.0 x ULN
* International normalized ratio (INR) =< 1.2
* Platelet (Plt) count > 30,000
* Ability to take oral medication (dasatinib must be swallowed whole)
* No clinically significant infections as determined by the investigator
* Normal corrected QT (QTc) interval (< 450 msec)
* Serum potassium and magnesium are within normal limits
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (sensitivity =< 25 IU HCG/L) within 72 hours prior to the start of study drug administration
* Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped prior to study enrollment; women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy
* After consent, discontinuation ("washout period") of any medications known to contribute significantly to the risk of QT prolongation or interfere with cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) mediated drug metabolism
* Patient agrees to discontinue St. John's Wort while receiving dasatinib therapy (discontinue St. John's Wort at least 5 days before starting dasatinib)
* Patient agrees that IV bisphosphonates will be withheld for the first eight weeks of dasatinib therapy due to risk of hypocalcemia
* Patient agrees to discontinue anti-coagulants and anti-platelet drugs; note: a low dose aspirin regimen (81mg QD) is permitted with close monitoring of the subject's platelets for a level >= 50,000/mm^3

Exclusion Criteria:

* Patients may not receive concurrent chemotherapy, radiotherapy, or immunotherapy
* Pleural or pericardial effusion of any grade
* Uncontrolled angina, > New York Heart Association (NYHA) class III congestive heart failure or myocardial infarction (MI) within 6 months prior to study enrollment
* Diagnosed congenital long QT syndrome
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
* Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
* Subjects who are detained or imprisoned are not eligible
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* May not take concomitant medications that are generally accepted to have a risk of causing Torsades de Pointes including: (patients must discontinue drug 7 days prior to starting dasatinib)

  * Quinidine, procainamide, disopyramide
  * Amiodarone, sotalol, ibutilide, dofetilide
  * Erythromycin, clarithromycin
  * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
  * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, sparfloxacin, lidoflazine
* Patients already taking other CYP inducers or inhibitors other than those listed above are eligible for the study only after principal investigator (PI) review; dose adjustments and/or monitoring of drug levels where applicable will be made as needed by the PI after consultation with pharmacy
* Women who:

  * Are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or
  * Have a positive pregnancy test at baseline, or
  * Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-10; Primary Completion 2016-07-12 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Spurgeon, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Dasatinib)
Started | 19
Completed | 13
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Dasatinib)
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With In Vitro Dasatinib Sensitivity in Predicting Clinical Activity
Description: Defined by a decrease in absolute lymphocyte count, as determined by peripheral blood complete blood count (CBC) with differential or by bone marrow examination of 50 % and/or a decrease of detectable total lymph node size or spleen size by 50% (either by clinical examination contrast enhanced computed tomography [CT]).
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Dasatinib)
Number analyzed (Participants) | 13
Participants
  In vitro dasatinib sensitivity in predicting clini | 5
  ABS lymph ct decrease > 50% | 4
  Total lymph size decrease > 50% | 4
  Spleen decrease by > 50% | 0
Statistical Analysis 1: Comparison: Treatment (Dasatinib); Percent change from baseline in responders compared to non-responders (lymph node size); Test type: Non-Inferiority — A non-parametric two-sided Mann-Whitney test was run assuming non-Gaussian distributions. Two-tailed with 95% confidence intervals; p = 0.0106, t-test, 2 sided; Threshold for statistical significance is 0.05
Statistical Analysis 2: Comparison: Treatment (Dasatinib); Percent change from baseline in responders compared to non-responders (Absolute Lymphocyte Count (ALC)); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.19860, t-test, 2 sided; Threshold for statistical significance is 0.05
Statistical Analysis 3: Comparison: Treatment (Dasatinib); Percent change from baseline in responders compared to non-responders (spleen size); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.5167, t-test, 2 sided; Threshold for statistical significance is 0.05

2. Secondary Outcome: Objective Response
Description: Proportion of patients achieving the endpoint along with its 95% exact binomial confidence interval will be presented. Complete Response (CR): present >=2 mos: no symptoms of CLL, normal findings on exam, ALC < 4.000/mm3, ANC >1.500/ mm3, platelet (PLT) count (ct) >100.000/ mm3, hemoglobin (Hgb) concentration >11 g/dL (untransfused), bone marrow (BM) lymphocytosis <30%, and no nodules (lymphoid aggregates) on BM biopsy. Partial Response (PR): present >=2 months: a reduction in prev. enlarged nodes, spleen, & liver by at least 50%. ANC >= 1.500/ mm3 or PLT ct >= 100.000/ mm3 or Hgb concentration >=11 g/dL or 50% improvement over pre-therapy reductions in Hgb concentration and/or PLT ct. Nodular PR: persistent BM nodules or infiltrates seen on BM biopsy those achieving a CR or PR. Stable Disease (SD): Does not meet CR or PR, but also not progressive disease (PD). PD: 50% size increase of lymph node, spleen, liver; or histologic (e.g. Richter's) transformation (per NCI and iwCLL).
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Dasatinib)
Number analyzed (Participants) | 13
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 2
  Partial Response with Lymphocytosis (PR-L) | 2
  Stable Disease (SD) | 8
  Progression | 1

3. Secondary Outcome: Overall Survival
Description: Kaplan-Meier method will be used to estimate the survival curve.
Time Frame: Up to 2 years
Population: Given the significant evolution of the treatment landscape, overall survival was no longer deemed to be a worthwhile/meaningful endpoint. Patients were lost to follow up and data was not collected.
Arm/Group | Treatment (Dasatinib)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier method will be used to estimate the survival curve.
Time Frame: Up to 2 years
Population: as for outcome 3
Arm/Group | Treatment (Dasatinib)
Number analyzed (Participants) | 0

5. Secondary Outcome: Incidence of Adverse Events (Number of Participants Affected)
Description: Assessed According to the NCI Common Terminology Criteria for Adverse Events Version 4.0. Adverse events will be tabulated and summarized according to key reporting criteria (i.e., grade or seriousness, unanticipated, treatment attribution). Refer to the Adverse Event tables below for specific details.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Dasatinib)
Number analyzed (Participants) | 13
Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected within 30 days of discontinuation of study drug, up to 4 years.
Description: Adverse events were tabulated and summarized according to key reporting criteria (i.e., grade or seriousness, unanticipated, treatment attribution).
Arm/Group | Treatment (Dasatinib)
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 8/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Dasatinib) (N=13)
Facial Swelling (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 3 Facial swelling
Colitis (Gastrointestinal disorders) | 1 (1) — Grade 3 Colitis
Fatigue (General disorders) | 2 (2) — Grade 3 Fatigue
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) — Grade 3 hypocalcemia
Edema (Blood and lymphatic system disorders) | 1 (1) — Grade 3 Edema
Bilateral leg edema (Blood and lymphatic system disorders) | 1 (1) — Grade 3 leg edema
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) — Grade 3 leukocytosis
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) — Grade 3 thrombocytopenia
Neutropenia (Blood and lymphatic system disorders) | 1 (1) — Grade 3 neutropenia
Anemia (Blood and lymphatic system disorders) | 2 (2) — Grade 3 Anemia
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1) — Grade 3 hyperkalemia
Conjunctivitis (Eye disorders) | 1 (1) — Grade 3 conjunctivitis
Pneumonia (Infections and infestations) | 1 (1) — Grade 3 organizing pneumonia
vasovagal reaction (General disorders) | 1 (1) — Grade 3 vasovagal reaction
basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 3 basal cell carcinoma

LIMITATIONS AND CAVEATS:
No limitations or caveats are noted at this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No